CLINICAL TRIAL: NCT00338403
Title: Effects of Continuous Airway Pressure on the Ability to Heat and Humidify Air
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 14357A
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: CPAP pressure of -5cm/water during cold, dry air exposure; CPAP pressure of 0cm/water during cold, dry air exposure; CPAP pressure of 5cm/water during cold, dry air exposure; CPAP pressure of 10cm/water during cold, dry air exposure
MeSH Terms: interventions — Continuous Positive Airway Pressure; Water

INTERVENTIONS:
Procedure: Continuous positive airway pressure (CPAP) at -5, 0, 5 and 10 cm of water

SUMMARY:
We hypothesize that continuous positive pressure applied to the airway will decrease the ability of the nose to warm and humidify inspired air compared to zero or negative pressure.

We will use continuous positive airway pressure (CPAP), a device commonly used to treat patients with sleep apnea, to vary the pressure in the airway and determine if increased pressure decreases the ability to warm and humidify inspired air. If our hypothesis is correct, it may explain the reason why CPAP is poorly tolerated in patients with sleep apnea; i.e., less ability to warm and humidify air leading to more nasal mucosal irritation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age.
2. A clinical history suggestive of normal nose and upper airway, other than during a cold.
3. Willingness of the subject to participate in and complete the study, and the ability to understand the purpose of the trial.

Exclusion Criteria:

1. Physical sign or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Women of childbearing potential who are pregnant, trying to become pregnant or nursing a child.
3. Subjects treated with systemic steroids during the previous 30 days.
4. Subjects treated with topical (inhaled, intranasal or intraocular) steroids, Nasalcrom or Opticrom during the previous 15 days.
5. Subjects treated with oral antihistamine/decongestants during the previous seven days.
6. Subjects treated with topical (intranasal or intraocular) antihistamine/decongestants during the previous 3 days.
7. Subjects treated with immunotherapy.
8. Subjects on chronic anti-asthma medications.
9. Subjects with polyps in the nose or a significantly displaced septum.
10. Subjects who have incurred an upper respiratory tract infection within 14 days of the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The amount of water evaporated during the last 5 minutes of exposure to cold, dry air

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Rouadi P, Baroody FM, Abbott D, Naureckas E, Solway J, Naclerio RM. A technique to measure the ability of the human nose to warm and humidify air. J Appl Physiol (1985). 1999 Jul;87(1):400-6. doi: 10.1152/jappl.1999.87.1.400. PMID 10409601
- [Result] Assanasen P, Baroody FM, Rouadi P, Naureckas E, Solway J, Naclerio RM. Ipratropium bromide increases the ability of the nose to warm and humidify air. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1031-7. doi: 10.1164/ajrccm.162.3.9912055. PMID 10988126
- [Result] Assanasen P, Baroody FM, Abbott DJ, Naureckas E, Solway J, Naclerio RM. Natural and induced allergic responses increase the ability of the nose to warm and humidify air. J Allergy Clin Immunol. 2000 Dec;106(6):1045-52. doi: 10.1067/mai.2000.110472. PMID 11112885
- [Result] Assanasen P, Baroody FM, Naureckas E, Solway J, Naclerio RM. The nasal passage of subjects with asthma has a decreased ability to warm and humidify inspired air. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1640-6. doi: 10.1164/ajrccm.164.9.2103086. PMID 11719303
- [Result] Assanasen P, Baroody FM, Naureckas E, Solway J, Naclerio RM. Supine position decreases the ability of the nose to warm and humidify air. J Appl Physiol (1985). 2001 Dec;91(6):2459-65. doi: 10.1152/jappl.2001.91.6.2459. PMID 11717205
- [Result] Pinto JM, Assanasen P, Baroody FM, Naureckas E, Solway J, Naclerio RM. Treatment of nasal inflammation decreases the ability of subjects with asthma to condition inspired air. Am J Respir Crit Care Med. 2004 Oct 15;170(8):863-9. doi: 10.1164/rccm.200309-1271OC. Epub 2004 Jun 1. PMID 15172894